CLINICAL TRIAL: NCT07146269
Title: Effectiveness of Virtual Reality-Based Relaxation as an Adjunctive Therapy to Optimize At-Home Transcranial Direct Current Stimulation (tDCS) for Depression: A Randomized Controlled Trial
Brief Title: Virtual Reality-Augmented At-Home tDCS for Major Depression
Acronym: VR-TMD
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Technical University of Munich (Other)
Responsible Party: Principal Investigator, Ulrike Vogelmann, Dr. med., Technical University of Munich
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RWNM_tDCS_VR
Record Dates: First submitted 2025-08-14; First posted 2025-08-28 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Major Depression Moderate; Major Depression Severe
Keywords: Non-invasive Brain Stimulation (NIBS); Major Depression; Virtual Reality (VR); Transcranial Direct Current Stimulation (tDCS); tDCS at-home
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tDCS only (Active Comparator): Transcranial Direct Current Stimulation (tDCS) at home, 20 sessions, 2mA (5 days/week, for 4 weeks)
  Interventions: Device: tDCS
- tDCS plus VR (Experimental): Transcranial Direct Current Stimulation (tDCS) at home plus Virtual Reality (VR)-based relaxation 20 sessions, 2mA (5 days/week, for 4 weeks)
  Interventions: Device: tDCS; Device: VR-based relaxation therapy

INTERVENTIONS:
Device: tDCS — Transcranial Direct Current Stimulation delivered at an intensity of 2 mA over electrodes at F3/F4 (bifrontal, over DLPFC), for 30 minutes a day, Monday to Friday, for a total 20 sessions.
Device: VR-based relaxation therapy — Nature exposure via a Virtual Reality (VR) headset, for 30 minutes daily concurrently to tDCS, Monday to Friday, for a total of 20 sessions.
  Arms: tDCS plus VR

SUMMARY:
The goal of this clinical trial is to investigate the efficacy of combining Virtual Reality (VR)-based relaxation and Transcranial Direct Current Stimulation (tDCS) for treating Major Depression.

The main questions this study aims to answer are:

1. Does the combination of VR Relaxation and tDCS at-home result in significantly greater symptom improvement in depression than tDCS alone?
2. Are there differences in treatment effectiveness depending on demographic characteristics (e.g., age, gender)?
3. Feasibility: What is the level of acceptance and adherence to the combined VR and tDCS therapy compared to tDCS alone?

In a randomized controlled trial, patients will be assigned to either a tDCS + VR group or a tDCS-only group.

The study protocol is the following:

* On the first day, patients complete baseline questionnaires and are then randomly assigned to either the tDCS-only group or the tDCS + VR group.
* Both groups perform home-based treatment five times per week for four weeks, with each session lasting 30 minutes.
* After two weeks, patients return for a follow-up visit to complete questionnaires and assess adherence, side effects, and clinical progress.
* At the end of the four-week treatment period, a final assessment is conducted, including questionnaires and patient feedback.
* After 12-16 weeks (i.e. 2 to 3 months after the last tDCS session) Follow Up Assessment (BDI, MADRS, HDRS, GCI, GAF)

DETAILED DESCRIPTION:
Participant Recruitment:

Patients with unipolar or bipolar depression will be recruited from inpatient wards at Klinikum rechts der Isar and outpatient services. After screening for eligibility and obtaining informed consent, participants will be randomized into two groups (1:1), stratified by depression severity (MADRS > or < 30):

Active Group: 4-week home-based combination therapy of tDCS and VR-based relaxation

Control Group: 4-week home-based tDCS without VR relaxation

Treatment Protocol:

at-home tDCS: 2 mA for 30 minutes, electrodes at F3/F4 (bifrontal, over DLPFC), daily Monday to Friday, total 20 sessions. Optional MRI before/after treatment.

VR Relaxation: Nature exposure via VR headset, 30 minutes daily parallel to tDCS, Monday to Friday, 20 sessions.

Assessment Schedule:

Baseline Visit (Visit 1): Informed Consent, demographics, medical history, vital signs, and baseline scales (BDI, MADRS, HDRS, GCI, GAF, CTQ, EHI, FTND). First session in-clinic with training for home use. Up to 5 additional sessions may be conducted in-clinic.

Mid-Treatment (Visit 2): After 2 weeks: vital signs, questionnaires (BDI, MADRS, HDRS, GCI, GAF), therapy adherence (according to number of conducted sessions), side effects, treatment adjustments if needed.

Final Assessment (Visit 3): After 4 weeks: final vitals, questionnaires (BDI, MADRS, HDRS, GCI, GAF), patient satisfaction survey, therapy experience interview.

Follow Up Assessment (Visit 4): After 12-16 weeks: questionnaires (BDI, MADRS, HDRS, GCI, GAF)

Technical data on tDCS use (automatic logging) including time, adherence, etc., will also be recorded.

ELIGIBILITY:
Inclusion Criteria:

* At least a moderate depressive episode (MADRS baseline score ≥ 20).
* Patients aged between 18 and 65 years.
* Sufficient cognitive abilities to understand study requirements and instructions (MMSE ≥ 27).
* Stable antidepressant/psychiatric medication for at least two weeks prior to study entry.

Exclusion Criteria:

* Currently clinically relevant Axis II disorders.
* Other relevant Axis I disorders (except anxiety disorders).
* Substance use disorders within the last 3 months prior to study entry (excluding nicotine and caffeine dependence).
* Skin lesions at the site of tDCS electrode placement.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-07-15 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Depressive symptoms assessed by MADRS | Measured at day 1 (baseline) and day 29 (after the full 4 weeks of treatment).
  Major Depression psychiatric symptoms assessed with the Montgomery Asberg Depression Rating Scale (MADRS). MADRS values are interpreted as follows: 0-6 = No depression, 07-19 = mild, 20-34 = moderate, 35-60 = severe.
  Primary outcome is the Difference in MADRS Score from baseline to post-treatment visit (day 29)

SECONDARY OUTCOMES:
Clinical Global Impression assessed by CGI-S | Measured at day 1 (baseline), day 15 (after 2 weeks of treatment), day 29 (after the full 4 weeks of treatment) and followup in 2-3 Months (after 12-16 weeks of treatment).
  Clinical Global Impression - Severity scale (CGI-S). Outcome values are interpreted as follows:
  1. - Normal, not at all ill
  2. - Borderline mentally ill
  3. - Mildly ill
  4. - Moderately ill
  5. - Markedly ill
  6. - Severely ill
  7. - Among the most extremely ill patients
Psychosocial functioning assessed by GAF score | Measured at day 1 (baseline), day 15 (after 2 weeks of treatment), day 29 (after the full 4 weeks of treatment) and followup in 2-3 Months (after 12-16 weeks of treatment).
  Global psychosocial functioning will be assessed using the Global Assessment of Functioning (GAF) scale. Outcome values are interpreted as follows:
  91-100 Excellent No symptoms; superior functioning 81-90 Good Minimal symptoms, generally doing well 71-80 Mild Some mild symptoms or difficulties 61-70 Moderate Mild symptoms but generally functioning 51-60 Moderate to serious Moderate symptoms or difficulty in functioning 41-50 Serious Serious symptoms or impairments 31-40 Major impairment Impairment in several areas (e.g., work, school) 21-30 Severe Behavior influenced by delusions, serious communication issues 11-20 Very severe Danger to self/others, gross communication issues 1-10 Extreme Persistent danger of severely hurting self/others 0 Not assessable Insufficient information
Depressive symptoms assessed by BDI-II | Measured at day 1 (baseline), day 15 (after 2 weeks of treatment), day 29 (after the full 4 weeks of treatment) and followup in 2-3 Months (after 12-16 weeks of treatment).
  Major Depression psychiatric symptoms assessed with the Beck Depression Inventory (BDI-II). Outcome values are interpreted as follows: 0-13 = Minimal depression, 14-19 = Mild depression, 20-28 = Moderate depression, 29-63 = Severe depression
Depressive symptoms assessed by HDRS | Measured at day 1 (baseline), day 15 (after 2 weeks of treatment), day 29 (after the full 4 weeks of treatment) and followup in 2-3 Months (after 12-16 weeks of treatment).
  Major Depression psychiatric symptoms assessed with the Hamilton Depression Rating Scale (HADRS). Outcome values are interpreted as follows: 0-7 = No Depression, 08-16 = mild, 17-23 = moderate, ≥ 24 = severe
Change in resting-state functional connectivity measured by resting-state fMRI (Fisher-z) between dorsolateral prefrontal cortex (DLPFC) and anterior cingulate cortex (ACC) in a subset of participants | Measured at day 1 (baseline) and day 29 (after the full 4 weeks of treatment).
  Resting-state fMRI-based Pearson correlation between average BOLD time series of DLPFC and ACC, computed per scanned participant and Fisher-z-transformed. Only participants who underwent fMRI are included.
  Measurement tool: Resting-state fMRI on 3T MRI scanner; ROI time-series extraction and correlation analysis Unit of measure: Fisher-z (dimensionless) How aggregated: Mean Fisher-z per participant; Change score = Day 29 - Day 1.
Change in resting-state functional connectivity measured by resting-state fMRI (Fisher-z) between anterior cingulate cortex (ACC) and amygdala | Measured at day 1 (baseline) and day 29 (after the full 4 weeks of treatment).
  Resting-state fMRI-based Pearson correlation between average BOLD time series of anterior cingulate cortex (ACC) and amygdala, Fisher-z-transformed.
  Measurement tool: Resting-state fMRI on 3T MRI scanner; ROI time-series extraction and correlation analysis.
  Unit of measure: Fisher-z (dimensionless) How aggregated: Mean Fisher-z per participant; Change score = Day 29 - Day 1.
Change in resting-state functional connectivity measured by resting-state fMRI (Fisher-z) between hippocampus and amygdala | Measured at day 1 (baseline), day 15 (after 2 weeks of treatment), and day 29 (after the full 4 weeks of treatment).
  Resting-state fMRI-based Pearson correlation between average BOLD time series of hippocampus and amygdala, Fisher-z-transformed.
  Measurement tool: Resting-state fMRI on 3T MRI scanner; ROI time-series extraction and correlation analysis.
  Unit of measure: Fisher-z (dimensionless) How aggregated: Mean Fisher-z per participant; Change score = Day 29 - Day 1.
Change in resting-state functional connectivity measured by resting-state fMRI (Fisher-z) between dorsolateral prefrontal cortex (DLPFC) and hippocampus | Measured at day 1 (baseline), day 15 (after 2 weeks of treatment), and day 29 (after the full 4 weeks of treatment).
  Resting-state fMRI-based Pearson correlation between average BOLD time series of dorsolateral prefrontal cortex (DLPFC) and hippocampus, Fisher-z-transformed.
  Measurement tool: Resting-state fMRI on 3T MRI scanner; ROI time-series extraction and correlation analysis.
  Unit of measure: Fisher-z (dimensionless) How aggregated: Mean Fisher-z per participant; Change score = Day 29 - Day 1.
Change in blood pressure (part of general physical health assessment) | Measured at day 1 (baseline), day 15 (after 2 weeks of treatment), and day 29 (after the full 4 weeks of treatment).
  Systolic blood pressure measured in mmHg. Values interpreted according to standard clinical reference ranges.
  Measurement tool: Standard sphygmomanometer or automated BP monitor Unit of measure: mmHg How aggregated: Mean systolic BP per participant; Change score = current day - baseline
Change in heart rate (part of general physical health assessment) | Day 1 (baseline), Day 15 (after 2 weeks of treatment), Day 29 (after 4 weeks of treatment)
  Description: Heart rate measured in beats per minute (bpm). Values interpreted according to standard clinical reference ranges.
  Measurement tool: Pulse oximeter, ECG, or manual measurement Unit of measure: beats per minute (bpm) How aggregated: Mean heart rate per participant; Change score = current day - baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- Technical University of Munich, TUM School of Medicine and Health, Department of Psychiatry and Psychotherapy, Munich, Germany

IPD SHARING:
Plan to Share IPD: Yes
All anonymised study outcomes will be shared, including questionnaire, physiological, and device data.
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: IPD and supporting information will be made available immediately after the publication of study results, for an unrestricted duration.
Access Criteria: The de-identified individual patient data, i.e., all IPD that underlie results in a publication, will be made accessible after its publication for non-commercial academic projects that have a legitimate research topic and a clearly stated hypothesis. In the event that the application is accepted, researchers will be asked to get the study approved by their institution's ethics board. The study principal investigator will subsequently provide the de-identified data sets via a safe data transfer system.